CLINICAL TRIAL: NCT01600001
Title: A Randomized, Double-blind, Placebo-controlled, Phase II Study of KWA-0711 in Patients With Chronic Idiopathic Constipation (CIC)
Brief Title: A Exploratory Study of KWA-0711 in Patients With Chronic Idiopathic Constipation (CIC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KWA1201
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Idiopathic Constipation
Keywords: Chronic Idiopathic Constipation (CIC); Constipation; Functional gastrointestinal disorders
MeSH Terms: conditions — Constipation; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Drug:KWA-0711 dose 1 (Experimental)
  Interventions: Drug: KWA-0711
- Drug:KWA-0711 dose 2 (Experimental)
  Interventions: Drug: KWA-0711
- Drug:KWA-0711 dose 3 (Experimental)
  Interventions: Drug: KWA-0711
- Drug:KWA-0711 dose 4 (Experimental)
  Interventions: Drug: KWA-0711
- Drug: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KWA-0711
  Arms: Drug:KWA-0711 dose 1; Drug:KWA-0711 dose 2; Drug:KWA-0711 dose 3; Drug:KWA-0711 dose 4
Drug: Placebo
  Arms: Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KWA-0711 in Chronic Idiopathic Constipation (CIC) patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients who experienced fewer than three SBMs per week for more than 6 months prior to the enrollment
* The patients who experienced one or more of the following signs or symptoms during more than 25% of bowel movements for more than 6 months: straining, lumpy or hard stools, and a sensation of incomplete evacuation

Exclusion Criteria:

* Patients who have secondary constipation caused by systemic disorder
* Patients who have organic constipation
* Patients who received intestinal resection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)

PRIMARY OUTCOMES:
Improvement of signs and symptoms associated with constipation | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Tokyo and Other Japanese City, Japan